CLINICAL TRIAL: NCT04024735
Title: Mechanisms of COPD Exacerbation Recurrence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 21022
Record Dates: First submitted 2019-04-04; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; COPD Exacerbation; Patient Readmission; Recurrence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Recurrence | interventions — Spirometry; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Spirometry, Forced Oscillation Technique, Step-counter, sputum and blood samples — We will be collecting demographic and clinical information including daily physical activity level, lung function, blood and sputum samples. These measurements will be collected at patient admission, discharge and at follow-up of 30 and 90 days.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common smoking-related lung disease. Patients with COPD are at increased risk of readmission to hospitals within the following 30 days. Hospital readmissions of COPD contribute to clinical and economic burden on society. Understanding why some COPD patients are readmitted remains a key area of unmet need.

To our knowledge, no previous study has fully investigated both the social and clinical risk factors associated with these types of patients. The investigators want to prospectively and comprehensively explore the possible causes, whether clinical or social factors, that cause rehospitalisation. The investigators will be collecting demographic and clinical information including daily physical activity level, lung function, blood and sputum samples. These measurements will be collected at patient admission, discharge and at follow-up of 30 and 90 days. This process could lead to a better understanding of the reasons which prevent early hospital readmission for those patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a primary diagnosis of COPD
* Patients admitted to hospital with an exacerbation.

Exclusion Criteria:

* Patients in whom an initial diagnosis of an AECOPD is revised to an alternative at a later phase of the study.
* Patients who have a predominant history of asthma
* Patients with a confirmed active malignancy
* Patients who have a predominant history of bronchiectasis.
* Cognitive impairment patients with a Mental Test Score (MTS) of 6 or less.
* Inability to give informed consent to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients admitted to the hospital because of COPD exacerbation.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the factors that determine readmission to hospital within 30 and 90 days post discharge. | 30 and 90 days

SECONDARY OUTCOMES:
Readmission rate at 30 days and at 3 months | 30 and 90 days
Prevalence of comorbidities between those who are and are not readmitted within 30 and 90 days. | 30 and 90 days
Changes in admission-to-discharge in within breath reactance (∆Xrs5Hz) between patients who are and are not readmitted to the hospital within 30 and 90 days. | 30 and 90 days
Change in the modified Medical Research Council scale (mMRC) at admission, discharge and after 30 days follow-up or at readmission. | 30 and 90 days
  It is used to scale breathlessness, ranges from 0 to 4 which higher values represent a worse outcome.
Change in quality of life by measuring COPD assessment test (CAT) at admission, discharge and after 30 days follow-up or at readmission. | 30 and 90 days
  It is used to scale patient's quality of life. Range of CAT scores from 0-40 which higher scores denote a more severe impact of COPD on a patient's life.
Change in Hospital Anxiety and Depression Scale (HADS) at admission, discharge and after 30 days follow-up or at readmission. | 30 and 90 days
  It is used to scale patient's quality of life. The questionnaire comprises seven questions for anxiety and seven questions for depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The higher score indicates a worse outcome.
Prevalence of frailty between those who are and are not readmitted to the hospital within 30 and 90 days. | 30 and 90 days
Change in physical activity level (daily steps) following the discharge between patients who are and are not readmitted. | 30 days
  Step counter (pedometer) will be given to wear throughout the 30 days period to measure the daily steps.
Changes in admission-to-discharge peak inspiration flow rate (PIFR) between patients who are and are not readmitted. | 30 and 90 days
  The In-Check DIAL device will be used which is capable of measuring inspiratory flow rates between 0 and 120 L/min. Optimal PIFR, more than 60 L/min; and sub-optimal PIFR, 60 L/min or less).
Change in white cell count (WCC) blood biomarkers | 30 and 90 days
  At admission, discharge and at readmission.
Change in C-reactive protein (CRP) blood biomarker | 30 and 90 days
  At admission, discharge and at readmission.
Change in Eosinophils blood biomarker | 30 and 90 days
  At admission, discharge and at readmission.
Change in Neutrophils blood biomarker | 30 and 90 days
  At admission, discharge and at readmission.
Change in troponin blood biomarker | 30 and 90 days
  At admission, discharge and at readmission.
Change in B-type Natriuretic Peptide (BNP) blood biomarker | 30 and 90 days
  At admission, discharge and at readmission.
Change in procalcitonin blood biomarker | 30 and 90 days
  At admission, discharge and at readmission.
Change in fibrinogen blood biomarker | 30 and 90 days
  At admission, discharge and at readmission.
Change in sputum biomarkers | 30 and 90 days
  This is used to assess bacteria species, load and resistance to antibiotics, and markers of inflammation such as IL-8.
Number of hospital admissions in the previous year. | 30 and 90 days
  The investigators will record it to find the difference between patients who are and are not readmitted to the hospital within 30 and 90 days.
Number of exacerbations in the previous year. | 30 and 90 days
  The investigators will record it to find the difference between patients who are and are not readmitted to the hospital within 30 and 90 days.
Use of long-term oxygen therapy (LTOT) | 30 and 90 days
  The investigators will record it to find the difference between patients who are and are not readmitted to the hospital within 30 and 90 days.
Length of stay (LOS) in hospital | 30 and 90 days
  The investigators will record it to find the difference between patients who are and are not readmitted to the hospital within 30 and 90 days.
Use of non-invasive ventilation (NIV) | 30 and 90 days
  The investigators will record it to find the difference between patients who are and are not readmitted to the hospital within 30 and 90 days.
Previous admission to the ICU | 30 and 90 days
  The investigators will record it to find the difference between patients who are and are not readmitted to the hospital within 30 and 90 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free Hospital NHS, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided